CLINICAL TRIAL: NCT00613691
Title: A Phase I, Open-label, Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the Endothelin B Agonist, SPI-1620, in Patients With Recurrent or Progressive Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-1620
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Carcinoma
Keywords: Refractory; Progressive
MeSH Terms: conditions — Carcinoma | interventions — sovateltide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPI-1620 (Experimental): SPI-1620 an endothelin B agonist
  Interventions: Drug: SPI-1620

INTERVENTIONS:
Drug: SPI-1620 — SPI-1620 in escalating doses from 0.5 μg/m2 intravenous over sixty seconds

SUMMARY:
This is a 2-part, open-label, single-arm, dose escalation study. Part I will define the Maximum Tolerated Dose (MTD) and optimal dose of SPI-1620 and evaluate its PK and PD properties. Once the MTD for SPI-1620 is identified, a second phase of the study will focus on dose escalation of docetaxel studied in groups of 3-6 patients. This part of the study will assess the safety and tolerability of increasing doses of docetaxel administered with the optimal dose of SPI 1620 defined in Part I.

DETAILED DESCRIPTION:
This is a 2-part, open-label, single-arm, dose escalation study. Part I will define the Maximum Tolerated Dose (MTD) and optimal dose of SPI-1620 and evaluate its PK and PD properties. Eligible patients will receive SPI-1620 delivered intravenously over one minute on Days 1, 8 and 15. On Day 8 patients will undergo a series of four H215O PET Blood Flow (BF) scans which will be used to assess alterations in BF induced by SPI-1620 in tumor and non-tumor ROIs (Region of Interest). Fifteen minutes after receiving SPI-1620 on Day 15, patients will receive docetaxel, 60 mg/m2, administered by infusion over 1 hour. Accelerated dose escalation of SPI-1620 will be employed: one patient will be treated at each dose level with 100% increases between dose levels. If any grade 2 or higher, related AE occurs, the trial will revert to 3-patient cohorts with 40% dose escalation between groups. There will be no intrapatient dose escalation. Dose escalation will continue until there is either no further increase in tumor blood flow as assessed by H215O PET scan, or until significant toxicity is observed. Once the MTD for SPI-1620 is identified, a second phase of the study will focus on dose escalation of docetaxel studied in groups of 3-6 patients. This part of the study will assess the safety and tolerability of increasing doses of docetaxel administered with the optimal dose of SPI 1620 defined in Part I. If 60 mg/m 2 was tolerated in Part I then up to six patients in Part II will receive docetaxel at a dose of 80 mg/m2 once every 3 weeks. If this is tolerated the next group of patients will receive docetaxel 100 mg/m2 once every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

All of the following inclusion criteria must be met prior to participation in this study

1. The patient must sign an informed consent. A signed consent form is required prior to the performance of any protocol-related procedures or assessments.
2. The patient must be >= 18 years of age.
3. The patient must have progressive or recurrent carcinoma and has failed all standard therapies for his/her tumor.
4. The patient must have a negative CT scan with contrast of the brain or MRI of the brain within 45 days of enrollment.
5. The patient must be using an acceptable/effective method of contraception if she is a female patient of childbearing potential.
6. The patient must have a negative serum pregnancy test within 14 days of entering the protocol if she is a female of childbearing potential.
7. The patient must have an ECOG score <= 2.
8. The patient must be willing and able to abide by the protocol.

Exclusion Criteria:

None of the exclusion criteria may be met prior to patient participation in this study

1. The patient has a history of CHF, migraines, coagulopathy, stroke or inadequately controlled hypertension.
2. The patient has asthma or symptomatic COPD.
3. The patient has autonomic nerve dysregulation syndrome.
4. The patient has angina or is taking nitrates or has had a MI within the past six months.
5. The patient has a significant ventricular arrhythmia, class III or IV CHF or has a known coronary stenoses >80% and has not undergone either angioplasty or CABG
6. The patient is taking phosphodiesterase inhibitors
7. The patient has malignant or poorly controlled hypertension (>160/100)
8. The patient has symptomatic orthostatic hypotension
9. The patient is taking arterial vasodilators such as nifedipine or amlodipine or alpha blockers such as terazosin, tamsulosin and prazosin.
10. The patient has a screening absolute neutrophil count less than 1.5 K/uL
11. The patient has a screening platelet count less than 100 K/uL.
12. The patient has a screening creatinine greater than 2.0 mg/dL
13. The patient has a screening amino alanine transferase (ALT), or aspartate aminotransferase (AST) > 2.5 times the upper limit of the laboratory reference range or a total bilirubin > 1.0 mg/dL.
14. The patient has a known immunodeficiency disorder.
15. The patient is enrolled, or the patient plans to enroll, in any concurrent study of another investigational product.
16. The patient is taking, or the patient is planning to take other cancer treatments during the study except for patients with prostate cancer using LHRH agonist therapy.
17. The patient has a known hypersensitivity to any of the components of SPI 1620 or to docetaxel.
18. The patient has previously failed treatment with docetaxel for his/her tumor and a dose of SPI-1620 that has been shown to enhance tumor blood flow has not been identified.
19. The patient does not have a tumor that is at least 1cm. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of SPI-1620 administered to patients with recurrent or progressive carcinoma who have failed all standard therapy. | every three weeks

SECONDARY OUTCOMES:
To assess the pharmacokinetic and pharmacodynamic profiles of SPI-1620 administered to patients with recurrent or progressive carcinoma who have failed all standard therapy. | one week
To identify the optimum dose of SPI-1620 to be used in future Phase II studies. | every three weeks
To assess the safety and tolerability of doses of docetaxel from 60 mg/m2 to 100 mg/m2 when given following infusion of SPI 1620. | every three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Tolcher, MD, Principal Investigator — START
Locations (1):
- START, San Antonio, Texas, United States